CLINICAL TRIAL: NCT04436029
Title: Descartes-11 Consolidation Treatment in Patients With High-Risk Multiple Myeloma Who Have Residual Disease After Induction Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cartesian Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC 11B
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Descartes 11 (Experimental)
  Interventions: Biological: Descartes 11

INTERVENTIONS:
Biological: Descartes 11 — Car T-cells

SUMMARY:
To assess Minimal Residual Disease (MRD)-negative Complete Response (sCR) rate after consolidation treatment with Descartes-11 in patients with high-risk myeloma who have residual disease following induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older at the time of enrollment
* High-risk multiple myeloma patients who complete pre-transplant induction treatment anti- myeloma drug combination (minimum 2 drugs).

Exclusion Criteria:

* Patients who are pregnant or lactating.
* Patients who have any active and uncontrolled infection. No blood cultures are necessary unless clinically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-04-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Stephenson Cancer Center Oklahoma University Health Science Centers, Oklahoma City, Oklahoma
  - Medical College of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Mohan M, Gundarlapalli S, Szabo A, Yarlagadda N, Kakadia S, Konda M, Jillella A, Fnu A, Ogunsesan Y, Yarlagadda L, Thalambedu N, Munawar H, Graziutti M, Al Hadidi S, Alapat D, Thanendrarajan S, Zangari M, van Rhee F, Schinke C. Tandem autologous stem cell transplantation in patients with persistent bone marrow minimal residual disease after first transplantation in multiple myeloma. Am J Hematol. 2022 Jun 1;97(6):E195-E198. doi: 10.1002/ajh.26530. Epub 2022 Mar 21. No abstract available. PMID 35285981
- [Derived] Mohan M, Hari P, Szabo A, Dhakal B, Chhabra S, D'Souza A. Long term follow up of newly diagnosed multiple myeloma patients treated with pembrolizumab consolidation post-autologous stem cell transplantation. Leuk Res. 2021 Oct;109:106648. doi: 10.1016/j.leukres.2021.106648. Epub 2021 Jun 23. No abstract available. PMID 34182226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from Feb to May 2021
Groups:
- Descartes 11: Descartes 11: CAR T cells
Period: Overall Study
Arm/Group | Descartes 11
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Descartes 11
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 70 [59 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3
  Turkey | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Stringent Complete Response
Description: Per IMWG 2016 Response Criteria Summary sCR: Complete response (CR) plus a normal free light chain ratio and no clonal cells in bone marrow (by immunohistochemistry). The FLC ratio must be Kappa/Lambda ≤ 4:1 or ≥ 1:2 after counting at least 100 plasma cells. CR: Negative immunofixation in serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow. VGPR: Serum M-protein detectable by immunofixation (not on electrophoresis) or a ≥ 90% reduction in M-protein, with urine M-protein <100 mg/24 hours. PR: ≥ 50% reduction in serum M-protein and a ≥ 90% reduction in 24-hour urinary M-protein (or to <200 mg/24 hours). If M-protein is unmeasurable, a ≥ 50% decrease in the difference between involved and uninvolved FLC levels is required. If both M-protein and serum-free light chains are unmeasurable, a ≥ 50% reduction in plasma cells is necessary, provided baseline plasma-cell percentage in bone marrow was ≥ 30%. Overall Response (OR): CR+VGPR+PR
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Descartes 11
Number analyzed (Participants) | 4
Participants | 1

ADVERSE EVENTS:
Time Frame: Through study completion, median follow up 6 months with a range of 1-9 months
Arm/Group | Descartes 11
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT04436029/Prot_SAP_002.pdf